CLINICAL TRIAL: NCT03563352
Title: Evaluating Nutritional Preferences and Product Accessibility in Oral Nutritional Supplements for Oncologic Patients - A Cross-Sectional Survey Study at Norris Comprehensive Cancer Center
Brief Title: Nutritional Preferences and Product Accessibility in Oral Nutritional Supplements in Participants With Breast, Colorectal, Upper Gastrointestinal, or Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Zero accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-17-4; NCI-2018-00948 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-17-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Breast Carcinoma; Cholangiocarcinoma; Colorectal Carcinoma; Gastric Carcinoma; Malignant Digestive System Neoplasm; Pancreatic Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview, survey): Participants attend an interview over 15 minutes and complete surveys.
  Interventions: Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Interview — Attend an interview
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies nutritional preferences and product accessibility in oral nutritional supplements in participants with breast, colorectal, upper gastrointestinal, or prostate cancer. Learning what participants like and dislike about their current or past used nutritional supplements may help doctor know how to improve them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify how patients with cancer are obtaining nutrition to support medical management.

SECONDARY OBJECTIVES:

I. Examine associations of gastrointestinal side effects with specific diagnoses and respective medical therapies.

II. Understand how patients access information regarding nutritional supplements.

III. Evaluate patient satisfaction with currently available oral nutritional supplements (ONS).

IV. Identify patient preferences in formulating a novel nutritional supplement.

OUTLINE:

Participants attend an interview over 15 minutes and complete surveys.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend English (both reading and writing)
* Subjects in the inpatient and outpatient setting with the diagnosis of breast cancer, colorectal cancer, upper gastrointestinal cancer (including gastric, pancreatic, and cholangiocarcinoma), or prostate cancer
* Receiving chemotherapy, biologic, or hormonal therapy in the University of Southern California (USC) Norris Comprehensive Cancer Center Day Hospital
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with a mental disability that makes them unable to understand and respond to the questions
* Patients with reported non-oncologic associated deficits in taste and smell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of breast cancer, colorectal cancer, upper gastrointestinal cancer (including gastric, pancreatic, and cholangiocarcinoma), and prostate cancer who are seen at the USC facilities will be screened and recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
The way patients with cancer choose and obtain nutritional supplements to support medical management | Up to 1 year
  Data from the oral nutritional supplement survey that examines quality, quantity, access and affordability of oral nutrional supplements will be summarized.

SECONDARY OUTCOMES:
Associations of gastrointestinal side effects with specific diagnoses and respective medical therapies | Up to 1 year
  Data from the survey will be used for testing the association of gastrointestinal side effects with specific diagnosis and medical therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States